CLINICAL TRIAL: NCT00779831
Title: Comparative, Randomized, Single Dose, 2 Way Crossover Bioavailability Study of Ranbaxy and Warner - Lambert (Sudafed ® 12 Hour) 120 mg Pseudoephedrine Hydrochloride Extended - Release Tablets in Healthy Adult Volunteers Under Fasting Conditions.
Brief Title: Bioequivalence Study on Pseudoephedrine HCl 120 mg ER Tablets Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AA16795
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence Pseudoephedrine hydrochloride 120 mg extended release tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 120 mg Pseudoephedrine hydrochloride extended release tablets of ranbaxy
  Interventions: Drug: 120 mg Pseudoephedrine hydrochloride extended release tablets
- 2 (Active Comparator): (Sudafed ® 12 hour) 120 mg Pseudoephedrine hydrochloride extended - release tablets
  Interventions: Drug: 120 mg Pseudoephedrine hydrochloride extended release tablets

INTERVENTIONS:
Drug: 120 mg Pseudoephedrine hydrochloride extended release tablets

SUMMARY:
Compare bioavailability of Pseudoephedrine hydrochloride extended release tablets (Ranbaxy Laboratories Limited) against reference product Sudafed ® 12-hour tablets 120 mg (Warner-Lambert) under fasting conditions.

DETAILED DESCRIPTION:
This was an open label, randomized, single dose, 2-way crossover, relative bioavailability study performed on a total of 36 healthy adult subjects (20 males and 16 females). Thirty five (35) subjects (19 males and 16 females) completed the clinical phase of the study. In each period, subjects were housed from at least 10 hours before dosing until after the 36 hour blood draw. Single oral 120 mg Pseudoephedrine hydrochloride doses were separated by a washout period of 7 days.

A total of thirty six (36) subjects (20 males and 16 females) were enrolled in the study. Out of which a total of thirty five (35) subjects (19 males and 16 females) completed the clinical phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* All subjects enrolled in this study met all inclusion and exclusion criteria, and were judged by the investigator to be normal, healthy volunteers

Subjects were included in the study if they met all of the following criteria:

1. Healthy adult male or female volunteers , 18 to 55 years of age
2. Weighing at least 52 kg for males and 45 kg for females and within 15% of their ideal weights (table of 'Desirable Weights of Adults', Metropolitan Life Insurance Company, 1983)
3. Medically healthy subjects with clinically normal laboratory profiles and ECGs
4. Females of child bearing potential should either be sexually inactive (abstinent) for 14 days prior to the first dose and throughout the study or be using one of the following acceptable birth control methods:

   1. Surgically sterile (bilateral tubal ligation, hysterectomy, bilateral oophorectomy) 6 months minimum
   2. IUD in place for at least 3 months
   3. Barrier methods (condom, diaphragm) with spermicide for at least 14 days prior to the first dose and throughout the study
   4. Surgical sterilization of the partner (vasectomy for 6 months minimum)
   5. Hormonal contraceptives for at least 3 months prior to the first dose of the study
   6. Other birth control methods may be deemed acceptable
5. Post menopausal women with amenorrhea for at least 2 years will be eligible
6. Voluntarily consent to participate in the study

Exclusion Criteria:

* Subjects were excluded from the study if there was evidence of any of the following at screening or at any time during the study:

  1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease
  2. In addition, history or presence of:

     1. Alcoholism or drug abuse within the past year
     2. Hypersensitivity or idiosyncratic reaction to Pseudoephedrine or any other sympathomimetic amines
     3. Glaucoma or hypermetropia
  3. Female subjects who are pregnant or lactating
  4. Positive results on HIV, HbsAg and HCV tests
  5. Subjects receiving a monoamine oxidase (MAO) inhibitor or within 14 days of stopping use of an MAO inhibitor, or any sympathomimetic amines
  6. Subjects who have been on a special diet (for whatever reason) during the 28 days prior to the first dose and throughout the study
  7. Subjects who through completion of the study, would have donated in excess of:
* 500 mL of blood in 14 days
* 1500 mL of blood in 180 days
* 2500 mL of blood in 1 year. 8. Subjects who have participated in another clinical trial within 28 days prior to the first dose.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2004-06; Primary Completion 2004-06 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- MDS Pharma Services, Saint-Laurent, Quebec, Canada

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html